CLINICAL TRIAL: NCT05575232
Title: Effectiveness and Usability of a Mobile Application to Assist in the Pharmacological and Non-pharmacological Treatment of Arterial Hypertension
Brief Title: Effectiveness and Usability of a Mobile Application to Assist in the Treatment of Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Aline Mendes Gerage, Principal investigator, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APP PRESSÃO NA BOA
Record Dates: First submitted 2022-09-13; First posted 2022-10-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: Hypertension; Mobile Health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application Group (GA) (Experimental): Participants undergoing the GA will be instructed on how to download the application and how to use it. From there, all personal data must be entered into the application so that alerts, tips and incentives can be issued to each one, individually.
  Interventions: Behavioral: Application Group (GA)
- Control Group (GC) (No Intervention): The GC, in turn, will participate in a single lecture, in the first week of the intervention, with basic guidelines related to the key points of the treatment of SAH, including the importance of medication adherence, monitoring of blood pressure values and/or capillary glucose, lifestyle modifications linked to physical activity, eating habits, smoking cessation, stress management and moderate alcohol consumption.

INTERVENTIONS:
Behavioral: Application Group (GA) — The main focus of the application is to assist in the treatment of patients with SAH. The application will address the components of adherence to medication use, blood pressure monitoring and promotion/monitoring of physical activity. In addition, health education tips will be provided, including guidelines for reducing sodium consumption, adopting an adequate and healthy diet, controlling body weight, moderate alcohol consumption and stress management, in accordance with the recommendations of the main guidelines related to the theme¹ ³. The intervention will last eight weeks.
  Arms: Application Group (GA)

SUMMARY:
Systemic arterial hypertension (SAH) is a multifactorial cardiovascular disease that stands out as an important risk factor for the development of other cardiovascular diseases, such as ischemic heart disease and stroke, which are the main causes of death in Brazil and in the world. In this sense, SAH is considered a major public health problem, given its high prevalence. However, despite the evidence of several effective treatments for SAH, in Brazil, it is estimated that 77% of hypertensive patients do not undergo any treatment. Among the possible reasons for this, the low adherence to the proposed treatment (pharmacological and non-pharmacological) and the deficiencies in health care systems in approaching the treatment of chronic diseases, such as SAH. In this context, in order to improve the control and treatment of patients with SAH, the development of innovative methodologies that provide strategies to increase adherence to drug treatment and facilitate changes in lifestyle are necessary. In this sense, the present proposal aims to develop an application for smartphones aimed at the treatment of SAH, with tools aimed at medication adherence, blood pressure monitoring, monitoring and promotion of physical activity and healthy lifestyle habits in hypertensive patients. Therefore, the study will be developed in three phases: Phase 1: application development; Phase 2: testing the effectiveness of the application in a controlled environment; and, Phase 3: usability testing of the application. In phase 2, a randomized controlled clinical trial will be conducted to test the effect of eight weeks of application use on laboratory blood pressure, physical activity level, adherence to medication treatment and general lifestyle. In Phase 3, the app will be available on Apple iTunes and Google Play. After the application is publicized in the media (advertisements on television, newspapers, radio) and in social groups, usability aspects will be evaluated, such as the number of downloads and the grade attributed to user evaluations, according to the sociodemographic characteristics of the user (sex, age, place of residence).

DETAILED DESCRIPTION:
The study will be developed in three stages, according to the objectives outlined. Initially, a prototype of a cellphone application will be developed to help Brazilian adults diagnosed with SAH, with tools related mainly to medication adherence, promotion of physical activity and monitoring of blood pressure values, in addition to health tips (food, smoking, alcoholism and stress management). Subsequently, this prototype will be made available to a group of adult hypertensive patients so that the effectiveness of this application can be tested on laboratory blood pressure values, medication adherence and lifestyle aspects, including physical activity and, subsequently, physical activity. Application usability will be tested. Subsequently, after making the necessary adjustments, the application will be made available on the Apple iTunes and Google Play platforms and disseminated in groups of Basic Health Units and in the media (advertisements on television, newspaper, radio). From there, the number of downloads and the grade assigned to user reviews (one, two, three or four stars) will be evaluated, according to the user's sociodemographic characteristics (gender, age, place of residence).

App Development

General Description

The main focus of the application is to assist in the treatment of patients with SAH. The application will address the components of adherence to medication use, blood pressure monitoring and promotion/monitoring of physical activity. In addition, health education tips will be provided, including guidelines for reducing sodium consumption, adopting an adequate and healthy diet, controlling body weight, moderate alcohol consumption and stress management, in accordance with the recommendations of the main guidelines related to the theme.

After downloading, patients must manually enter demographic data (date of birth, sex), their body mass and height, information regarding the use of the drugs used, the presence of comorbidities (diabetes, dyslipidemia, chronic kidney disease, coronary artery disease, peripheral arterial disease, among others). In addition, the user must enter data related to their lifestyle, including information about: physical activity, nutrition, alcohol consumption, tobacco use, stress and relationships, according to an adapted version of the Fantastic lifestyle.

Based on this information entered by the patient (input), the application will issue reminders: a) for the use of the medication(s), according to the time registered by the patient, daily; b) to perform blood pressure measurements. The patient will be instructed to take blood pressure measurements while sitting, in a calm environment, after five minutes of rest, with the bladder emptied and there is at least 30 minutes of abstention from food, cigarettes and/or alcoholic and caffeinated beverages. Such measured BP values must be entered in the application and, if a BP level above the recommended values is identified, the insertion of the importance of the correct use of antihypertensive medication and adoption of a healthy lifestyle will increase. It will also be suggested that you consult your doctor for possible medication adjustments.

In addition, the user will be given the possibility to self-monitor their physical activities and, based on this information, the application will generate feedback informing whether or not the user has reached the recommendations currently in force. If the user does not meet the recommendations throughout the week, illustrative messages or videos will be generated with stimuli and guidelines for the patient to increase their level of physical activity, according to such recommendations. Illustrative messages or educational videos will also be made available with tips on healthy living habits, including recommendations for body weight control, reducing sodium consumption, adopting healthy eating habits, stress control and smoking cessation, as recommended by the main guidelines related to thematic.

Reports for the patient regarding blood pressure values and physical activity will be available, showing the evolution over time. For programmers and researchers, these same reports will also be generated, in addition to reports with application usage statistics and general user characteristics (business intelligence), so that, with this information, the system can be feedback.

Patients will be able to designate family members and/or friends to have access to the data captured and generated by the application, so that these people can provide social support for the treatment of hypertensive patients. In addition, a communication channel will be opened between patients that the application identifies in closer locations, in case the patient wants to share doubts, challenges and achievements.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of SAH;
* Have been using antihypertensive medication for more than three months;
* Cannot be involved in the regular practice of physical activities.
* Have a smartphone.
* Not have cognitive disabilities that limit the understanding and use of an application and/or physical limitations that make it difficult to practice physical activities;

Exclusion Criteria:

* Changes in the type and/or dose of antihypertensive drugs used during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in clinic systolic blood pressure | up to 8 weeks
  The laboratory blood pressure (systolic and diastolic) will be obtained in two days, at a similar time, using the OMRON automatic equipment, model 742HEM. On each day, three measurements will be performed with an interval of one minute between them, with the cuff placed on the left arm, elevated to the height of the midpoint of the sternum. If the variation of these three measurements is greater than 4 mmHg for systolic and/or diastolic blood pressure, new measurements will be performed until this established criterion is met. The average value between the measurements obtained on the different days will be recorded as a reference value at the different moments of the study.
Changes in clinic diastolic blood pressure | up to 8 weeks
  The laboratory blood pressure (systolic and diastolic) will be obtained in two days, at a similar time, using the OMRON automatic equipment, model 742HEM. On each day, three measurements will be performed with an interval of one minute between them, with the cuff placed on the left arm, elevated to the height of the midpoint of the sternum. If the variation of these three measurements is greater than 4 mmHg for systolic and/or diastolic blood pressure, new measurements will be performed until this established criterion is met. The average value between the measurements obtained on the different days will be recorded as a reference value at the different moments of the study.

SECONDARY OUTCOMES:
Changes in medication adherence levels | up to 8 weeks
  Will be assessed using the Morisky's Therapeutic Adherence Scale of eight items
Changes in physical activity leves | up to 8 weeks
  Will be assessed using accelerometry, using devices of the GT3X and GT3X+ models (Actigraph Pensacola, FL, USA) and the Actilife software (Actigraph Pensacola, FL, USA)
Changes in lifestyle | up to 8 weeks
  Will be evaluated using an adapted version of the Fantastic questionnaire which includes questions related to the following components: nutrition, physical activity, preventive behavior, social relationships and stress control. For each question, patients will answer whether such behavior is not part of their lifestyle, rarely matches, almost always matches, or always matches.
Patient satisfaction with the application | through study completion, an average of 8 weeks
  Patients undergoing the GA will be invited to answer an adapted version of the assessment scale for smartphone applications for health care, proposed by Jim and Kim 24, which contains 23 items in total, related to the assessment of content, objectivity, interface design, writing style and technology, with response options ranging from zero (not at all) to four (a lot), generating an overall score.

CONTACTS AND LOCATIONS:
Overall Officials: ALINE M GERAGE, PHD, Study Chair — UNIVERSIDADE FEDERAL DE SANTA CATARINA (UFSC)
Locations (1):
- Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F, Redon J, Dominiczak A, Narkiewicz K, Nilsson PM, Burnier M, Viigimaa M, Ambrosioni E, Caufield M, Coca A, Olsen MH, Schmieder RE, Tsioufis C, van de Borne P, Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S, Clement DL, Coca A, Gillebert TC, Tendera M, Rosei EA, Ambrosioni E, Anker SD, Bauersachs J, Hitij JB, Caulfield M, De Buyzere M, De Geest S, Derumeaux GA, Erdine S, Farsang C, Funck-Brentano C, Gerc V, Germano G, Gielen S, Haller H, Hoes AW, Jordan J, Kahan T, Komajda M, Lovic D, Mahrholdt H, Olsen MH, Ostergren J, Parati G, Perk J, Polonia J, Popescu BA, Reiner Z, Ryden L, Sirenko Y, Stanton A, Struijker-Boudier H, Tsioufis C, van de Borne P, Vlachopoulos C, Volpe M, Wood DA. 2013 ESH/ESC guidelines for the management of arterial hypertension: the Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). Eur Heart J. 2013 Jul;34(28):2159-219. doi: 10.1093/eurheartj/eht151. Epub 2013 Jun 14. No abstract available. PMID 23771844
- [Background] Sociedade Brasileira de Cardiologia; Sociedade Brasileira de Hipertensao; Sociedade Brasileira de Nefrologia. [VI Brazilian Guidelines on Hypertension]. Arq Bras Cardiol. 2010 Jul;95(1 Suppl):1-51. No abstract available. Portuguese. PMID 21085756
- [Background] Barroso WKS, Rodrigues CIS, Bortolotto LA, Mota-Gomes MA, Brandao AA, Feitosa ADM, Machado CA, Poli-de-Figueiredo CE, Amodeo C, Mion Junior D, Barbosa ECD, Nobre F, Guimaraes ICB, Vilela-Martin JF, Yugar-Toledo JC, Magalhaes MEC, Neves MFT, Jardim PCBV, Miranda RD, Povoa RMDS, Fuchs SC, Alessi A, Lucena AJG, Avezum A, Sousa ALL, Pio-Abreu A, Sposito AC, Pierin AMG, Paiva AMG, Spinelli ACS, Nogueira ADR, Dinamarco N, Eibel B, Forjaz CLM, Zanini CRO, Souza CB, Souza DDSM, Nilson EAF, Costa EFA, Freitas EV, Duarte EDR, Muxfeldt ES, Lima Junior E, Campana EMG, Cesarino EJ, Marques F, Argenta F, Consolim-Colombo FM, Baptista FS, Almeida FA, Borelli FAO, Fuchs FD, Plavnik FL, Salles GF, Feitosa GS, Silva GVD, Guerra GM, Moreno Junior H, Finimundi HC, Back IC, Oliveira Filho JB, Gemelli JR, Mill JG, Ribeiro JM, Lotaif LAD, Costa LSD, Magalhaes LBNC, Drager LF, Martin LC, Scala LCN, Almeida MQ, Gowdak MMG, Klein MRST, Malachias MVB, Kuschnir MCC, Pinheiro ME, Borba MHE, Moreira Filho O, Passarelli Junior O, Coelho OR, Vitorino PVO, Ribeiro Junior RM, Esporcatte R, Franco R, Pedrosa R, Mulinari RA, Paula RB, Okawa RTP, Rosa RF, Amaral SLD, Ferreira-Filho SR, Kaiser SE, Jardim TSV, Guimaraes V, Koch VH, Oigman W, Nadruz W. Brazilian Guidelines of Hypertension - 2020. Arq Bras Cardiol. 2021 Mar;116(3):516-658. doi: 10.36660/abc.20201238. No abstract available. English, Portuguese. PMID 33909761
- [Background] Mansur Ade P, Favarato D. Mortality due to cardiovascular diseases in Brazil and in the metropolitan region of Sao Paulo: a 2011 update. Arq Bras Cardiol. 2012 Aug;99(2):755-61. doi: 10.1590/s0066-782x2012005000061. Epub 2012 Jun 28. English, Portuguese. PMID 22735870
- [Background] Azambuja MI, Foppa M, Maranhao MF, Achutti AC. Economic burden of severe cardiovascular diseases in Brazil: an estimate based on secondary data. Arq Bras Cardiol. 2008 Sep;91(3):148-55, 163-71. doi: 10.1590/s0066-782x2008001500005. English, Portuguese. PMID 18853056
- [Background] Uhlig K, Patel K, Ip S, Kitsios GD, Balk EM. Self-measured blood pressure monitoring in the management of hypertension: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 6;159(3):185-94. doi: 10.7326/0003-4819-159-3-201308060-00008. PMID 23922064
- [Background] Clark NM. Management of chronic disease by patients. Annu Rev Public Health. 2003;24:289-313. doi: 10.1146/annurev.publhealth.24.100901.141021. Epub 2001 Nov 6. PMID 12415147
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Marcolino MS, Oliveira JAQ, D'Agostino M, Ribeiro AL, Alkmim MBM, Novillo-Ortiz D. The Impact of mHealth Interventions: Systematic Review of Systematic Reviews. JMIR Mhealth Uhealth. 2018 Jan 17;6(1):e23. doi: 10.2196/mhealth.8873. PMID 29343463
- [Background] Palmer MJ, Barnard S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2018 Jun 22;6(6):CD012675. doi: 10.1002/14651858.CD012675.pub2. PMID 29932455
- [Background] Morawski K, Ghazinouri R, Krumme A, Lauffenburger JC, Lu Z, Durfee E, Oley L, Lee J, Mohta N, Haff N, Juusola JL, Choudhry NK. Association of a Smartphone Application With Medication Adherence and Blood Pressure Control: The MedISAFE-BP Randomized Clinical Trial. JAMA Intern Med. 2018 Jun 1;178(6):802-809. doi: 10.1001/jamainternmed.2018.0447. PMID 29710289
- [Background] Mohammadi R, Ayatolahi Tafti M, Hoveidamanesh S, Ghanavati R, Pournik O. Reflection on Mobile Applications for Blood Pressure Management: A Systematic Review on Potential Effects and Initiatives. Stud Health Technol Inform. 2018;247:306-310. PMID 29677972
- [Background] Brazilian Institute of Geography and Statistics. Continuous National Household Sample Survey, Rio de Janeiro, 2017.
- [Background] Dayer LE, Shilling R, Van Valkenburg M, Martin BC, Gubbins PO, Hadden K, Heldenbrand S. Assessing the Medication Adherence App Marketplace From the Health Professional and Consumer Vantage Points. JMIR Mhealth Uhealth. 2017 Apr 19;5(4):e45. doi: 10.2196/mhealth.6582. PMID 28428169
- [Background] Muller AM, Alley S, Schoeppe S, Vandelanotte C. The effectiveness of e-& mHealth interventions to promote physical activity and healthy diets in developing countries: A systematic review. Int J Behav Nutr Phys Act. 2016 Oct 10;13(1):109. doi: 10.1186/s12966-016-0434-2. PMID 27724911
- [Background] Kumar N, Khunger M, Gupta A, Garg N. A content analysis of smartphone-based applications for hypertension management. J Am Soc Hypertens. 2015 Feb;9(2):130-6. doi: 10.1016/j.jash.2014.12.001. Epub 2014 Dec 11. PMID 25660364
- [Background] Tudor-Locke C, Craig CL, Brown WJ, Clemes SA, De Cocker K, Giles-Corti B, Hatano Y, Inoue S, Matsudo SM, Mutrie N, Oppert JM, Rowe DA, Schmidt MD, Schofield GM, Spence JC, Teixeira PJ, Tully MA, Blair SN. How many steps/day are enough? For adults. Int J Behav Nutr Phys Act. 2011 Jul 28;8:79. doi: 10.1186/1479-5868-8-79. PMID 21798015
- [Background] Physical Activity Guidelines Advisory Committee. 2018 Physical Activity Guidelines Advisory Committee Scientific Report. Washington, DC: US Department of Health and Human Services, 2018.
- [Background] Gerage AM, Benedetti TRB, Cavalcante BR, Farah BQ, Ritti-Dias RM. Efficacy of a behavior change program on cardiovascular parameters in patients with hypertension: a randomized controlled trial. Einstein (Sao Paulo). 2020 Jan 31;18:eAO5227. doi: 10.31744/einstein_journal/2020AO5227. eCollection 2020. PMID 32022106
- [Background] Oliveira-Filho AD, Barreto-Filho JA, Neves SJ, Lyra Junior DP. Association between the 8-item Morisky Medication Adherence Scale (MMAS-8) and blood pressure control. Arq Bras Cardiol. 2012 Jul;99(1):649-58. doi: 10.1590/s0066-782x2012005000053. Epub 2012 Jun 7. English, Portuguese. PMID 22688844
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Jin M, Kim J. Development and Evaluation of an Evaluation Tool for Healthcare Smartphone Applications. Telemed J E Health. 2015 Oct;21(10):831-7. doi: 10.1089/tmj.2014.0151. Epub 2015 Jun 4. PMID 26431261

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT05575232/Prot_SAP_ICF_000.pdf